CLINICAL TRIAL: NCT05986643
Title: Using Biofeedback During Exergaming to Attenuate Alpha Oscillations to Improve Postural Control in People Living With Parkinson's.
Brief Title: Brain Training to Improve Balance in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: University of Exeter (Other); University of Nottingham (Other); University of Plymouth (Other); European Bioinformatics Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0903; 324686 (Other: HRA)
Record Dates: First submitted 2023-04-19; First posted 2023-08-14 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: Balance; Gait
MeSH Terms: conditions — Parkinson Disease | interventions — Exergaming; Single Person

STUDY DESIGN:
Intervention Model Description: To maintain the gold standard approach of complete randomisation but we have tightened the inclusion criteria to stipulate both a history of falls and freezing of gait (FoG).
Who Masked: Investigator
Masking Description: Random computer generation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergame & Neurofeedback (Active Comparator): Six 5 minutes sets of participants standing on a balance board within virtual environment playing the exergame and receiving real neurofeedback with 1 minute rest between each set.
  Interventions: Behavioral: Exergame+Neurofeedback
- Exergame & SHAM Feedback (Sham Comparator): Six 5 minutes sets of participants standing on a balance board within virtual environment playing the exergame and receiving SHAM neurofeedback with 1 minute rest between each set.
  Interventions: Behavioral: Exergame [alone]

INTERVENTIONS:
Behavioral: Exergame+Neurofeedback — Electroencephalography (EEG) is a device that measures the electrical activity of the brain (brain waves). There are several frequencies of brain waves when we are awake; alpha (medium), beta (fast), and theta (slow). Alpha frequencies of brain activity are linked to maintaining balance, with more alpha activity being associated with poorer balance. EEG neurofeedback treatment involves placing electrodes on a person's head to monitor and change brain activity by giving cued audio or visual feedback. It has been used in PwP to show improvements in balance and walking. Other preliminary research in PwP has shown that exercise can also improve balance.
  Arms: Exergame & Neurofeedback
Behavioral: Exergame [alone] — The exergame, delivered in virtual reality, involves travelling down a road (to give optic flow) whilst dodging balls that move towards the participant by either shifting their body either to the left or right. They are also be instructed to stand still and catch stars that appear and these will be used to score points and are associated with a monetary reward, ensuring motivation.
  This group will receive SHAM feedback.
  Other Names: Exergame
  Arms: Exergame & SHAM Feedback

SUMMARY:
People living with Parkinson's (PwP) rank balance problems amongst the most disabling symptom. Over time, balance function continues to decline and PwP go on to fall, affecting between 45-68% of PwP. Falling directly impacts upon the individuals' quality of life (QoL), as it prevents patients from doing everyday activities, and places PwP at greater risk of other medical problems, such as fractures.

New treatments are urgently needed to improve balance and reduce falls in order to improve QoL for PwP. The aim of this project is to achieve these goals by using exercise to alter brain activity. Supporting our idea, are previous studies that show both exercise alone as well as changing brain activity at rest via visual feedback (similar to how breathing can be controlled to lower blood pressure), can be used to rehabilitate balance. Here researchers test the idea that better results can be achieved for PwP, if a specific exercise program is used as the feedback to change brain activity.

PwP will be assigned randomly into 2 groups, one receiving the exergaming physical therapy (PT) alone with a placebo feedback and, the second group will be required to change brain activity using exercise feedback to change brain activity.

Each intervention will be performed 3 times/week with each session lasting 1⁄2 an hour, for 12 consecutive weeks. Participants are expected to attend 5 sessions over each fortnight. Assessments of balance will be made before and after all three treatments. This will allow us to measure any improvements and compare the 2 different methods to see which one improves balance the most in PwP.

DETAILED DESCRIPTION:
This is a multi-centre centre study with University of Leicester and DeMontfort University being research sites. NHS organisations will be PIC sites where participants will be identified from. No medical data or access to patient medical records will be made. A PIC mNCA will be in place with NHS organisations.

For the design of the study, the investigators will adopt a double-blinded randomised clinical trial. This means that patients will not know their group allocation and the research associate that will be analysing the data will also not know what treatment the patient received.

Participants will be allocated into either group 1 or 2. Participants in both groups will both perform the exergame rehabilitation. The exergame, delivered in virtual reality, involves travelling down a road (to give optic flow) whilst dodging balls that move towards the participant by either shifting their body either to the left or right. Patients are also be instructed to stand still and catch stars that appear, and these will be used to score points and are associated with reward, ensuring motivation.

This exergame has been specifically designed to combine aspects of movement and balance control, body position, aerobic fitness, strengthening of core muscles and elements of co-ordination and speed.

The difference between the two groups will be the neuro-feedback provided during the performance of the exercise game. That is, group 1 will receive real feedback of brain activity whilst group 2 will receive a placebo which is called SHAM feedback. This corresponds to a random recording that has no association/correlation with on-going brain (EEG) activity. All participants will be randomly assigned a unique key code via a random computer generator, this will be facilitated by the Data Monitoring and Ethics committee. The research technician, that will perform the analysis of the data, will not be privy to particular intervention of interest. After the random allocation, but before the intervention, all participants will receive a familiarisation procedure for their allocation. Once the participants have successfully undergone the eligibility screening (see section below for details), participants will be randomly allocated to one of two groups. The research team will then conduct the familiarisation sessions before proceeding to the pre-intervention assessment (limit of stability at baseline). This will be followed by the 12-week training program (that requires attendance at 30 1/2hr sessions over the course of three months. This will be followed by the 12 week (end of program) post-intervention assessment to measure the limit of stability, and a further single follow-up at 6 months to asses for long-term retention of any benefits. The 12-week post-intervention testing sessions will occur within 72 hours, but no less than 24 hours following the preceding training session. For the Pre-and Post- assessments: this will include the : (i) the Limits of Stability test, (ii) Sensory Organisation Test, (iii) Parkinson's Disease Questionnaire, (iv) Berg Balance Scale, (v) Section III of UPDRS, (vi) mBEST, (vii) 6 Metre WalkTest, (viii) 4 Square Step Test, and (ix) the Daily Activities Questionnaire. All of the aforementioned measures are openly available and do not require any licenses/permission to use. Accordingly, there will not be any need to share data with the license holders.

VISIT 1:

In the first visit the research team will firstly ensure that the PLwP meet the eligibility criteria and that none of the exclusion criteria apply. Only those eligible will be randomly allocated to one or two groups, and the research team will measure using posturography and walking assessments to obtain a baseline balance score. The research team will also complete questionnaires, including the Parkinson's Disease Questionnaire, Berg Balance Scale, Section III of the UPDRS, and Daily Activities Questionnaires. The research team will also take a brief medical history. This initial visit will take place at the balance testing laboratory at DeMonfort University.

12 WEEK TRAINING PROGRAMME: During the 12-week training programme, participants will be asked to attend the balance laboratory at the University of Leicester, where either the exergame activity with feedback from brain activity or no feedback will be performed. These training sessions will last half an hour in total, and it is expected patients to complete 5 sessions over the course of a 2- week period. An online booking system will be used to manage the sessions. Participants will be allowed to miss a total of 6 sessions in total across the whole of the 3-month intervention program. Missing any more that this would compromise the integrity of the data.

POST INTERVENTION:

A post-intervention will be arranged immediately at the end of the training programme, then again at 3 and 6 months respectively. During these post-interventions, measurements will be taken from using the posturography and walking assessments to obtain a baseline balance score. Questionnaires will be completed, including the Parkinson's Disease Questionnaire, Berg Balance Scale, Section III of the UPDRS, and Daily Activities Questionnaires. A brief medical history will be taken again. These visits will take place at the balance testing laboratory at DeMonfort University.

INTERVIEWFor the optional part of the study, an interview will be arranged to take the patients' and Carers views on the accessibility and tolerability of these interventions, these will take place roughly 2 weeks at the end of the final training session. An encrypted voice recorder will be used. Participant ID will be mentioned at the beginning of the recording so that participants remain anonymous. Recordings will be stored in a secure environment at the University before the recordings are transferred to university computers. Recordings will be immediately deleted as soon as the recordings have been transferred. The research team or an external transcribing company (a confidentiality agree will be in place), will transcribe the recordings for analysing.

ELIGIBILITY:
Inclusion Criteria:

People with Parkinson with mild-moderate disease and severe disability (but able to stand and walk unaided (Hoehn and Yahr stage ≤4) be eligible if:

* in everyday life, they do less than the recommended aerobic exercise for older adults (i.e., vigorous exercise done <3 times per week, 20 min per session; or moderate exercise done <5 times per week, 30 min per session).
* they have experienced at least one fall and one episode of freezing of gait in the past year.
* they are taking stable dopaminergic pharmacotherapy (stable dose for at least 1 month) or are still without treatment and not expected to start treatment within the next 3 months.

As long as all criteria are met - we will not impose any lower (assuming they are adults) or upper age limit for recruitment.

Exclusion Criteria:

* severe lower limb motor impairments and/or requirement of a walking aid or wheelchair
* previously diagnosed with stroke or dementia
* having metal implants in the head (i.e. deep brain stimulator or aneurysm clips)
* any other known medical, mental health, or physical condition which may interfere with balance.
* patients on beta-blocking agents or antipsychotics
* patients with other neurological, orthopaedic, or cardiac co-morbidities that make them unfit to do exercise or interferes with balance and cognitive functions required to participate in this study
* patients with psychiatric diseases diagnosed in the past year by a psychiatrist
* patients with dementia
* those unable to tolerate the exergame task.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-04 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Balance Scores | 12 weeks
  Changes in balance scores using The Limits of stability (LOS) test. This dynamic balance score is measured using a commercially available system (Bertec CDP/IVRTM (Interacoustics)).The participants will be asked to stand barefoot on the centre of the force platform, and will be support by a secure harness throughout to prevent falls. The assessment requires each participant to move their centre of pressure (COP) towards an intended target in the following order: forward, forward right, right, backward right, backward, backward left, left and forward left. Movement velocity (degrees per second), maximal excursion (greatest distance [cm] achieved towards the intended target/maximal distance of target [cm]) and directional control ([the amount of intended movement - amount of extraneous movement)/amount of intended movement] × 100) will be measured, representing the maximum distance an individual can intentionally sway without losing balance or needing to take a step.

SECONDARY OUTCOMES:
Sensory Organisation Scores | 12 weeks
  Changes in the Sensory Organisation test scores, calculated by an interval scale, with 100 indicating no sway and 0 indicating an uncompleted trial.
  This task comprises six different sensory conditions in quiet stance and measures the COP path in centimetres. The test progressively becomes harder by either distracting or removing visual and/or proprioceptive feedback. During sway-referenced conditions, erroneous sensory information is presented to the participant while the force platform measures the participant's ability to compensate by using other senses to maintain balance. The following sensory conditions will be used:
  * Condition 1: Eyes open and fixed support
  * Condition 2: Eyes closed and fixed support
  * Condition 3: Eyes open sway-referenced and support sway-referenced
  * Condition 4: Eyes open and support sway referenced
  * Condition 5: Eyes closed and support sway-referenced
  * Condition 6: Eyes open and sway-referenced with support sway-referenced
Daily Life Scores | 12 weeks
  Changes of activities in daily life.
  The investigators will use a validated questionnaire to asses functional improvements in activities associated with everyday living.
  Activities of Daily Living Questionnaire (ADLQ) - A questionnaire aimed for use with patients diagnosed with cognitive impairments, which assesses function in ADL tasks across 6 areas of life.
  A set of four descriptions of different competence levels; scores range from 0 to 3 where higher scores indicate greater impairment. A fifth response option, "don't know/has never done" is also available, and if this option is selected, the item is excluded from scoring.

CONTACTS AND LOCATIONS:
Overall Officials: Qadeer Arshad, Principal Investigator — University of Leicester
Locations (1):
- University of Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
We plan to share via open access platforms the study protocol and statistical analysis approach before commencing the trial.
Supporting Information: Study Protocol, SAP
Time Frame: Before the trial commences
Access Criteria: No criteria

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-10-09): https://cdn.clinicaltrials.gov/large-docs/43/NCT05986643/SAP_000.pdf